CLINICAL TRIAL: NCT06184321
Title: A Randomized Trial of Alteplase Versus Placebo Through an Indwelling Pleural Catheter for Management of Symptomatic Septated MPE
Brief Title: Alteplase Through an Indwelling Pleural Catheter for the Management of Symptomatic Septated Malignant Pleural Effusion
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0554; NCI-2021-09122 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0554 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (alteplase) (Experimental): Patients receive alteplase instilled into the IPC which is capped for 1-2 hours before the catheter is drained.
  Interventions: Biological: Alteplase
- Arm II (placebo) (Placebo Comparator): Patients receive placebo instilled into the IPC which is capped for 1-2 hours before the catheter is drained. Beginning 1 week later, patients may receive alteplase as in arm I.
  Interventions: Drug: Placebo Administration

INTERVENTIONS:
Biological: Alteplase — Instilled into IPC
  Other Names: Activase; Plasminogen Activator (Human Tissue-Type Protein Moiety); r-tPA; Recombinant Tissue Plasminogen Activator; rt-PA
  Arms: Arm I (alteplase)
Drug: Placebo Administration — Instilled into IPC
  Arms: Arm II (placebo)

SUMMARY:
This study investigates whether alteplase can help to improve pleural fluid drainage and dyspnea (breathlessness) in patients with non-draining malignant pleural effusion. Alteplase helps dissolve blood clots and is used to treat heart attacks, strokes, and clots in the lungs. Alteplase may help to control symptoms of breathlessness.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate dyspnea using the visual analog scale (VAS) scale at one week in patients with symptomatic septated malignant neoplasm of the pleural effusion (MPE) and a non-draining/inadequately draining indwelling pleural catheter (IPC).

SECONDARY OBJECTIVE:

I. To evaluate dyspnea using the visual analog scale (VAS) scale at 48 hours (+/-12 hours) after treatment with intrapleural alteplase, in patients with septated MPE and a nondraining/inadequately draining IPC. In addition, complications, quality adjusted survival (calculated using the SF-6D to determine utilities and then integrating utilities over time to arrive at quality-adjusted survival), change in dyspnea (using the Borg score and VAS scale) at 1 week (+/- 1 day), 2 weeks (+/- 2 days) and every 4 weeks (+/- 2 days) after the intervention until IPC removal or death.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive alteplase instilled into the IPC which is capped for 1-2 hours before the catheter is drained.

ARM II: Patients receive placebo instilled into the IPC which is capped for 1-2 hours before the catheter is drained. Beginning 1 week later, patients may receive alteplase as in arm I.

ELIGIBILITY:
Inclusion Criteria:

* Referral to pulmonary services for inability to drain fully via IPC
* Presence of a symptomatic septated pleural effusion
* A pleural effusion of significant moderate to large volume based on:

  * Chest radiograph: effusion filling >= 1/3 of the hemithorax, or
  * Computed tomography (CT)-scan: AP depth of the effusion >= 1/3 of the AP dimension on the axial image superior to the hemidiaphragm, including atelectatic lung surrounded by effusion, or
  * Ultrasound: effusion spanning at least three intercostal spaces, with a >= 3 cm in at least one intercostal space, while the patient sits upright
* Age > 18
* Borg score >= 3
* Absence of a blocked IPC as demonstrated by a flush with 20 cc of saline x1 without resistance
* Presence of septated effusion based on ultrasound (US) and chest CT

Exclusion Criteria:

* Inability to provide informed consent
* Study subject has any disease or condition that interferes with safe completion of the study including:

  * Uncorrectable coagulopathy based on criteria followed by cardiopulmonary center for procedures.
  * Active bleeding
  * Known allergic reaction to thrombolytics
* Pleural effusion is smaller than expected on bedside pre-procedure ultrasound
* No septations and/or no loculations on bedside pre-procedure ultrasound
* Patient is asymptomatic
* Blocked IPC as determined by saline flush

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Horiana Grosu, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org